CLINICAL TRIAL: NCT03547622
Title: Pilot Study of Galantamine and CBT4CBT to Reduce Post-taper Relapse for MAT
Brief Title: Galantamine and CBT4CBT Pilot to Prevent Relapse.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000021868; 2P50DA009241-21 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-06-06 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: Methadone or Buprenorphine Detoxoxification
MeSH Terms: interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAT taper with galantamine (Active Comparator): Following initial MAT taper, participants will be given up to 16mg daily of galantamine for up to 10 weeks of the active study
  Interventions: Drug: MAT taper with galantamine
- MAT taper with placebo (Placebo Comparator): Following initial MAT taper, participants will be given up to 16mg daily of placebo for up to 10 weeks of the active study
  Interventions: Drug: MAT taper with placebo

INTERVENTIONS:
Drug: MAT taper with galantamine — Following taper from MAT (methadone or buprenorphine) participants will be given galantamine daily with access to a CBT4CBT computer program
  Other Names: Razadyne ER, Razadyne
  Arms: MAT taper with galantamine
Drug: MAT taper with placebo — Following taper from MAT (methadone or buprenorphine) participants will be given placebo daily with access to a CBT4CBT computer program
  Arms: MAT taper with placebo

SUMMARY:
The investigators are proposing a randomized pilot feasibility study to evaluate the effects of galantamine versus placebo on preventing relapse to opioid use following tapering from methadone or buprenorphine maintenance (Medication Assisted Treatment, or MAT) among adults with opioid use disorder, with additional behavioral therapy (web-based cognitive behavioral therapy) provided across all conditions to help individuals successfully transition from MAT to a drug-free state.

DETAILED DESCRIPTION:
This is a randomized pilot study to examine the potential use of galantamine as an adjunct to the standard buprenorphine or methadone taper in the context of behavioral support. Early abstinence from opioids is associated with high relapse rates and there is a great need to develop interventions that will prevent relapse to opioid use.

In this randomized pilot, 30 adults enrolled in the methadone or buprenorphine maintenance programs at the APT Foundation and who have sought a medically supervised, voluntary taper from these medications will be offered participation in a double-blind, placebo controlled, randomized trial of galantamine as an adjunct to standard tapering procedures at this clinic along with the combined approach utilizing concurrent behavior therapy. Primary outcomes will be: (1) successful completion of taper (achieving a methadone/buprenorphine dose of 0), (2) opioid withdrawal symptoms, and (3) opioid use, assessed by self-report and urine samples during and up to 3 months after the end of opioid taper. The investigators will also closely monitor patient comfort and safety (assessed by opioid withdrawal symptoms, adverse events, with measures of stress, sleep and pain) as well as cognitive function (assessed by the CANTAB).

ELIGIBILITY:
Inclusion Criteria:

* Are male and females, between the ages of 18 and 65
* Are enrolled in the APT methadone or buprenorphine program, have been stabilized for at least one year, and who voluntarily wish to taper off MAT.
* For women of child-bearing age, have a negative serum pregnancy test at screening, agree to adequate contraception to prevent pregnancy, and agree to have monthly urine pregnancy tests at the clinic.
* Are fluent in English and have a 6th grade or higher reading level.
* Can commit to at least 12 weeks of treatment and are willing to be randomized to treatment

Exclusion Criteria:

* Are undergoing administrative (non-voluntary) tapering (e.g., example due to non-payment of program fees, program rule infractions).
* Meet DSM-V psychiatric classifications for lifetime schizophrenia or bipolar disorder, or have a depressive or anxiety disorder with current use of a prescribed psychotropic medication that cannot be discontinued;
* Current DSM-V diagnosis of drug or alcohol use disorder (other than opioids or tobacco);
* Demonstrate significant medical conditions, including asthma or chronic obstructive lung disease, history or current gastrointestinal ulcer, hepatic or renal impairment and cardiac rhythm disturbances or any other medical conditions that the study physician deems contraindicated for galantamine treatment;
* Use of other medications including a) drugs that slow heart rate (e.g., beta-blockers),which may increase the risk of bradycardia and AV block and b) NSAIDs; increased potential for developing ulcers/active or occult gastrointestinal bleeding;
* Have a screening liver function test (AST or ALT) greater than 3 times normal;
* Known allergy or adverse reaction to galantamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Carroll, PhD, Principal Investigator — Yale University
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MAT Taper With Galantamine | MAT Taper With Placebo
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAT Taper With Galantamine | MAT Taper With Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (19.7) | 48.3 (17.6) | 43.8 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Medication dose-Methadone [Mean (Standard Deviation); unit: mg] — Population: Participants could be taking either Methadone or Buprenorphine for the study and dose in mg differs for the two medications.
  mg
    number analyzed (Participants) | 1 | 2 | 3
    (all) | 20 | 13.0 (1.4) | 15.3 (4.1)
Medication dose-Buprenorphine [Mean (Standard Deviation); unit: mg] — Population: Participants could be taking either Methadone or Buprenorphine for the study and dose in mg differs for the two medications.
  mg
    number analyzed (Participants) | 2 | 1 | 3
    (all) | 2.5 (2.1) | 2.0 | 2.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Methadone/Buprenorphine Dose to 0 mg for Successful Completion of Taper
Description: Number of participants who were able to taper to 0 mg from methadone or buprenorphine over 10 weeks of treatment.
  Data about current medication and dose in mg was collected at the start of treatment (week 1) was recorded on a weekly medical sheet. Data was then collected weekly from participant self-report and verified through the clinic database.
Time Frame: during 10 weeks of study and up to 3 months after the end of opioid taper
Measure: Count of Participants; unit: Participants
Arm/Group | MAT Taper With Galantamine | MAT Taper With Placebo
Number analyzed (Participants) | 3 | 3
Participants | 3 | 2

2. Secondary Outcome: Clinical Opioid Withdrawal Scale (COWS)
Description: opioid withdrawal score at week 0 (baseline) and at 10 weeks (post treatment).
  11-item scale designed to be administered by a clinician. Rates common signs and symptoms of opiate withdrawal and can be monitored over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. Score of 5-12 = mild; 13-24=moderate; 25-36=moderately severe; more than 36=severe withdrawal (Scale of 0 to 40).
Time Frame: Data at week 0 (baseline) and week 10 (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAT Taper With Galantamine | MAT Taper With Placebo
Number analyzed (Participants) | 3 | 3
score on a scale
  Week 0 (baseline) Score | 0 (0) | .33 (.58)
  Week 10 (Post Treatment Score) | 4.3 (5.1) | 4.2 (4.1)

3. Secondary Outcome: Substance Use Calendar
Description: number of days of opioid use, assessed by self-report
Time Frame: during 10 weeks of study
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MAT Taper With Galantamine | MAT Taper With Placebo
Number analyzed (Participants) | 3 | 3
Days | 1.0 (1.73) | 0 (0)

ADVERSE EVENTS:
Time Frame: 10 weeks of taper
Arm/Group | MAT Taper With Galantamine | MAT Taper With Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03547622/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03547622/ICF_001.pdf